CLINICAL TRIAL: NCT03376334
Title: A Pilot Study to Investigate the Effect of Motor Imagery on Dynamic Balance of Asymptomatic University Students: An Experimental Study
Brief Title: A Pilot Study to Investigate the Effect of Motor Imagery on Dynamic Balance of Asymptomatic Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Pramod Divakara Shenoy, MPT, Mr, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U/SERC/40/2014
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Balance
Keywords: Mental motor imagery; SEBT

STUDY DESIGN:
Intervention Model Description: One group received Mental Motor Imagery training, and the other group acted as a control with no specific intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor (using balance test) was not aware of neither the group to which the subject belonged nor to the baseline values of the subjects' balance score
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor Imagery (MI) (Experimental): Those meeting the inclusion criteria were selected (n=22). Each participant was necessary to complete the Movement Imagery Questionnaire in a quiet room. Finally, each participant assigned a score by using a 7-point scale regarding the ease/difficulty associated with representing each movement mentally. Next their baseline balance measurement was performed using the SEBT. Later this group had 9 motor imagery sessions, each session for 15 minutes, 3 sessions (alternate days) per week for a total of 3 weeks. Reassessment of balance was done after every 3 sessions.
  Interventions: Other: Mental Motor Imagery
- Control (C) (No Intervention): Those meeting the inclusion criteria were selected (n=10). Baseline measurement of SEBT was done on day 1, end of week 1, end of week 2 and end of week 3.

INTERVENTIONS:
Other: Mental Motor Imagery
  Arms: Motor Imagery (MI)

SUMMARY:
This study intended to investigate the effect of imagining a movement task on dynamic balance of sedentary university students. Two groups with good mental imaging ability were studied; one group receiving instructions on mental imagery and the other served as a control receiving no particular intervention. Any improvement in the balance ability was measured using the star excursion balance test (SEBT); for it has good to excellent test-retest reliability and validity as established by several researchers.

DETAILED DESCRIPTION:
Motor imagery (MI) refers to a cognitive process during which the representation of a specific motor action is internally simulated without producing an overt body movement. Motor imagery is now widely used as a technique to enhance motor learning and to enhance recovery during rehabilitation of various conditions such as sports injuries, stroke, etc. Several studies have also shown improvement in strength, function, and use of both upper and lower extremities in chronic stroke. Present study aimed to identify its effectiveness in improving dynamic balance of individuals without any clinical problem. Such improvement, if any, may be useful in early balance and proprioceptive training during the maximum protection phase of joint injuries, fractures, or even rehabilitation of other clinical conditions affecting balance. It may have benefits in maintaining / improving movements in athletes after injuries as well as the general less active population, including the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* No prior involvement in any physical or mental balance training
* Good mental imaging ability as determined using the motor imagery questionnaire

Exclusion Criteria:

* neuromusculoskeletal condition that may alter balance
* vestibular disorders or VBA related disorders
* painful conditions of the body
* H/o seizure, schizophrenia, meningitis, migraine, diplopia, spinal injuries, lower extremity injuries

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10-02 (Actual); Primary Completion 2015-05-25 (Actual); Study Completion 2015-05-25 (Actual)

PRIMARY OUTCOMES:
Dynamic Balance | 24 days
  Ability to balance while performing a task i.e. lower limb reach distance is various directions measured using star excursion balance test

SECONDARY OUTCOMES:
Time for improvement in balance | 7 to 24 days
  Time required to observe a significant improvement in balance

CONTACTS AND LOCATIONS:
Overall Officials: PRAMOD D SHENOY, MPT, Principal Investigator — Universiti Tunku Abdul Rahman; Yee Mun Chang, Principal Investigator — Alumnus of Universiti Tunku Abdul Rahman
Locations (1):
- Universiti Tunku Abdul Rahman, Cheras, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hosseini SA, Fallahpour M, Sayadi M, Gharib M, Haghgoo H. The impact of mental practice on stroke patients' postural balance. J Neurol Sci. 2012 Nov 15;322(1-2):263-7. doi: 10.1016/j.jns.2012.07.030. Epub 2012 Aug 1. PMID 22857987